CLINICAL TRIAL: NCT01213537
Title: A Study of the Effect of Cardiac Resynchronisation Therapy (CRT) on Chemosensitivity in Patients With Chronic Heart Failure With and Without Sleep Disordered Breathing.
Brief Title: Cardiac Resynchronisation Study
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Principal Investigator, Rebecca Lucas, Mrs, Imperial College London
Other Study IDs: 10/H0706/5
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Heart Failure
Keywords: Heart failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing clinically indicated CRT implantation: Patients may be included in the study if they fulfil the following;
  1. Age ≥18 years old
  2. Fulfil the current guidance for the implantation of a CRT device; optimal medical treatment for heart failure, broad QRS complex on electrocardiogram with or without evidence of cardiac dyssynchrony as appropriate, LVEF <35%, functional impairment as defined by an NYHA class of III-IV
  3. Clinically stable with no unplanned admission to hospital for preceding 4 weeks
  4. No changes in medications for heart failure in preceding 4 weeks
  5. Able to read and understand patient information sheet and give informed consent
  Patients must be excluded from the study if they fulfil they the following;
  1. On positive pressure treatment for known sleep disordered breathing at the time of inclusion
  2. Other known condition (untreated) likely to significantly disturb sleep eg. Restless legs syndrome, pain from any cause etc.
  3. Pregnancy

SUMMARY:
This study aims to investigate the effect of a pacemaker device used in heart failure patients which is called Cardiac Resynchronisation Therapy (CRT). Specifically the investigators aim to investigate if the CRT pacemaker has an effect on breathing stability in these patients and particularly breathing stability at night. Our theory is that the CRT pacemaker may improve the stability of breathing in patients with heart failure.

DETAILED DESCRIPTION:
AIM To investigate the effect of Cardiac Resynchronisation Therapy (CRT) on chemosensitivity in patients with Chronic Heart Failure with and without Sleep Disordered Breathing (SDB).

OBJECTIVE To conduct a physiological observational study to measure hypercapnic ventilatory responses in a group of CHF patients before and 3 months after implantation of clinically indicated CRT devices. Additionally to conduct nocturnal polysomnography to establish if any change in chemosensitivity is related to the presence of SDB at baseline and, where present, any change in SDB after implantation.

HYPOTHESIS Primary hypothesis: CRT implantation will be associated with a reduction in the hypercapnic ventilatory response from baseline to 3 months post implantation.

Additional hypothesis: This reduction in hypercapnic ventilatory response after CRT implantation will be greatest in those CHF patients with SDB at baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Fulfil the current guidance for the implantation of a CRT device; optimal medical treatment for heart failure, broad QRS complex on electrocardiogram with or without evidence of cardiac dyssynchrony as appropriate, LVEF <35%, functional impairment as defined by an NYHA class of III-IV
3. Clinically stable with no unplanned admission to hospital for preceding 4 weeks
4. No changes in medications for heart failure in preceding 4 weeks
5. Able to read and understand patient information sheet and give informed consent

Exclusion Criteria:

1. On positive pressure treatment for known sleep disordered breathing at the time of inclusion
2. Other known condition (untreated) likely to significantly disturb sleep eg. Restless legs syndrome, pain from any cause etc.
3. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Heart Failure who fulfil the current national guidelines for CRT insertion (see inclusion criteria)
Sampling Method: Probability Sample
Enrollment: 182 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change in chemosensitivity before and after CRT implantation | 3 months
  We will look primarily at the effect of CRT implantation on chemosensitity which we will measure using the ventilatory sensitivity to carbon dioxide.

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Brompton Hospital, London, London, United Kingdom

REFERENCES:
- See also: National Institute of Clinical Excellence; technology appraisal about CRT devices — http://www.nice.org.uk/TA120